CLINICAL TRIAL: NCT04347733
Title: Additive Effects of Hyaluronidase in Intra-articular Steroid Injection Treating the Initial Stage of Adhesive Capsulitis for Shoulder
Brief Title: Hyaluronidase in Intra-articular Steroid Injection Treating the Adhesive Capsulitis for Shoulder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Veterans Health Service Medical Center, Seoul, Korea (Other)
Responsible Party: Principal Investigator, Wonjae Lee, MD PhD, Director for the department of physical medicine and rehabilitation, Veterans Health Service Medical Center, Seoul, Korea
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-03-011-001
Record Dates: First submitted 2020-04-09; First posted 2020-04-15 (Actual); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Adhesive Capsulitis of Shoulder
Keywords: Intra-articular injections; Steroids; Hyaluronidase; Ultrasonography
MeSH Terms: conditions — Bursitis | interventions — Triamcinolone Acetonide; Hyaluronoglucosaminidase

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): Intra-articular injection, 20 mg (0.5 mL) of triamcinolone acetonide mixed with 2 mL of 2% lidocaine and 7.5 mL of normal saline
  Interventions: Drug: Triamcinolone Acetonide 40mg/mL
- Group B (Experimental): 40 mg (1 mL) of triamcinolone acetonide mixed with 2 mL of 2% lidocaine and 7.0 mL of normal saline
  Interventions: Drug: Triamcinolone Acetonide 40mg/mL
- Group C (Active Comparator): 20 mg (0.5 mL) of triamcinolone acetonide and 1 mL of hyaluronidase mixed with 2 mL of 2% lidocaine and 6.5 mL of normal saline
  Interventions: Drug: Triamcinolone Acetonide 40mg/mL; Drug: Hyaluronidase Injection

INTERVENTIONS:
Drug: Triamcinolone Acetonide 40mg/mL — We aimed to examine the therapeutic efficacy of the combination of hyaluronidase and steroid injection for adhesive capsulitis and to determine whether such a combination therapy might enable the total amount of steroids to be reduced.
Drug: Hyaluronidase Injection — We aimed to examine the therapeutic efficacy of the combination of hyaluronidase and steroid injection for adhesive capsulitis and to determine whether such a combination therapy might enable the total amount of steroids to be reduced.
  Other Names: Hirax Inj® BMI KOREA Pharmaceutical, South Korea
  Arms: Group C

SUMMARY:
Adhesive capsulitis (AC) is painful and disabling condition that is associated with a gradual loss of shoulder motion. Intra-articular steroid injection is a common treatment in the initial painful stage of AC, and its use in combination with hyaluronidase may offer increased therapeutic efficacy owing to synergistic effects. We determined the therapeutic efficiency of the co-administration of hyaluronidase in early AC by evaluating symptomatic, anthropometric, and imaging changes.

DETAILED DESCRIPTION:
We enrolled eligible patients with primary adhesive capsulitis in the initial stage.The subjects were randomly assigned into 3 groups to receive ultrasound-guided intra-articular injections with 20 mg (group A) and 40 mg triamcinolone acetonide (group B) and 20 mg acetonide combined with hyaluronidase (group C). The outcome measures included the visual analogue scale (VAS), the shoulder disability questionnaire (SDQ), abduction and external rotation range of motion, and intra-sheath fluid (ISF) before treatment and at 2, 4, 8, and 16 weeks after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Normal findings on simple x-rays of the shoulder but limitations in passive range of motion on physical examination
* Increased intra-sheath fluid (ISF) sufficient to encircle the long head of the biceps tendon within the upper portion of the bicipital groove of the humerus.

Exclusion Criteria:

* Ultrasonographic diagnosis of other concomitant fundamental abnormalities causing shoulder pain such as rotator cuff tear, bicipital tendon rupture, calcific tendinopathy, and subacromial-subdeltoid bursitis
* A history of shoulder injury
* A history of more than 1 year of conservative treatment for chronic shoulder pain
* Corticosteroid or hyaluronidase injections within the prior 6 months
* Hemiplegic shoulder
* Self-reported history consistent with scapula fracture or disarticulation
* Ipsilaterally cervical herniated intervertebral disc or brachial plexus injury
* Diabetes mellitus refractory to insulin therapy or glycated hemoglobin greater than 6.5
* Refusal to participate in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2019-03-27 (Actual); Study Completion 2019-07-16 (Actual)

PRIMARY OUTCOMES:
Change of visual analogue scale (VAS) | Evaluation at 5 time intervals: before injection and at 2, 4, 8, and 16 weeks after the injection
  Evaluation for the change of VAS that means average degree of shoulder pain for 24 hours before the evaluation (from 0 to 10 points)

SECONDARY OUTCOMES:
Change of shoulder disability questionnaire (SDQ) | Evaluation at 5 time intervals: before injection and at 2, 4, 8, and 16 weeks after the injection
  Evaluation for the change of SDQ that means the self-reported functional status in patients with shoulder disorders, comprised of 16 questions, reflecting the pain during various movements related with activities of daily living, with scores ranging from 0 (no disability) to 16 (greatest possible disability).
Change of degree for the abduction motion of shoulder | Evaluation at 5 time intervals: before injection and at 2, 4, 8, and 16 weeks after the injection
  Evaluation for the change of degree for the motion of shoulder, checked with an inclinometer, as a passive maneuver, in the supine position
Change of degree for the flexion motion of shoulder | Evaluation at 5 time intervals: before injection and at 2, 4, 8, and 16 weeks after the injection
  Evaluation for the change of degree for the motion of shoulder, checked with an inclinometer, as a passive maneuver, in the supine position
Change of area for the intra-sheath fluid | Evaluation at 5 time intervals: before injection and at 2, 4, 8, and 16 weeks after the injection
  Evaluation for the change of area for the intra-sheath fluid, checked and calculated ultrasonographically at the upper portion of the bicipital groove of the humerus.

CONTACTS AND LOCATIONS:
Overall Officials: Wonjae Lee, MD, Ph D, Study Director — Veterans Health Service Medical Center, Seoul, Korea
Locations (1):
- Veterans Health Service Medical Center, Seoul, South Korea

REFERENCES:
- [Background] Fields BKK, Skalski MR, Patel DB, White EA, Tomasian A, Gross JS, Matcuk GR Jr. Adhesive capsulitis: review of imaging findings, pathophysiology, clinical presentation, and treatment options. Skeletal Radiol. 2019 Aug;48(8):1171-1184. doi: 10.1007/s00256-018-3139-6. Epub 2019 Jan 3. PMID 30607455
- [Background] Ahn JH, Lee DH, Kang H, Lee MY, Kang DR, Yoon SH. Early Intra-articular Corticosteroid Injection Improves Pain and Function in Adhesive Capsulitis of the Shoulder: 1-Year Retrospective Longitudinal Study. PM R. 2018 Jan;10(1):19-27. doi: 10.1016/j.pmrj.2017.06.004. Epub 2017 Jun 12. PMID 28619380
- [Background] Tandon A, Dewan S, Bhatt S, Jain AK, Kumari R. Sonography in diagnosis of adhesive capsulitis of the shoulder: a case-control study. J Ultrasound. 2017 Aug 21;20(3):227-236. doi: 10.1007/s40477-017-0262-5. eCollection 2017 Sep. PMID 28900523
- [Background] Byun SD, Park DH, Hong YH, Lee ZI. The additive effects of hyaluronidase in subacromial bursa injections administered to patients with peri-articular shoulder disorder. Ann Rehabil Med. 2012 Feb;36(1):105-11. doi: 10.5535/arm.2012.36.1.105. Epub 2012 Feb 29. PMID 22506242
- [Result] Buhren BA, Schrumpf H, Hoff NP, Bolke E, Hilton S, Gerber PA. Hyaluronidase: from clinical applications to molecular and cellular mechanisms. Eur J Med Res. 2016 Feb 13;21:5. doi: 10.1186/s40001-016-0201-5. PMID 26873038
- [Result] Cho CH, Song KS, Kim BS, Kim DH, Lho YM. Biological Aspect of Pathophysiology for Frozen Shoulder. Biomed Res Int. 2018 May 24;2018:7274517. doi: 10.1155/2018/7274517. eCollection 2018. PMID 29992159